CLINICAL TRIAL: NCT06401018
Title: Comparison of the Effects of Music and Ambient Noise Cancelling on Post-operative Pain, Anxiety and Functional Outcome During Total Knee Arthroplasty.
Brief Title: Comparison of Music and Ambient Noise Cancellation in Patients Undergoing Total Knee Arthroplasty (TKA)
Acronym: TKA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Güzelali Özdemir, Professor, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: TABED 1-24-81
Record Dates: First submitted 2024-03-29; First posted 2024-05-06 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Knee Osteoarthritis; Anxiety; Post Operative Pain; Noise Exposure
Keywords: Total Knee Arthroplasty; Knee Replacement Surgery; Knee Osteoarthritis; Noise Cancelling; Ambient Noise; Post Operative Pain; Anxiety
MeSH Terms: conditions — Osteoarthritis, Knee; Anxiety Disorders; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: In our study, the patient population was divided into three groups according to the type of exposure to ambient noise during surgery.
Who Masked: Outcomes Assessor
Masking Description: The investigator who evaluates the trial will not know which method has been used on which patient, and will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Patients who do not undergo noise cancellation during surgery (Active Comparator): Patients who do not undergo noise cancellation during knee replacement surgery
  Interventions: Procedure: No noise cancellation and no music playing
- Patients undergoing noise cancellation during surgery (Active Comparator): Patients undergoing noise cancellation with the help of an over the head earmuff with noise cancelling properties during knee replacement surgery
  Interventions: Procedure: Noise cancelled but not allowed to listen to music
- Patients who were played music during the operation (Active Comparator): Patients who were played music that has been shown to reduce anxiety during surgery.
  Interventions: Procedure: Music is played but noise is not cancelled

INTERVENTIONS:
Procedure: No noise cancellation and no music playing — In this group of patients, no apparatus was used to prevent noise in the environment, and they were not exposed to any music in the environment.
  Arms: Patients who do not undergo noise cancellation during surgery
Procedure: Noise cancelled but not allowed to listen to music — In this group of patients, only noise cancelling was performed during the operation, but no music was played in the environment.
  Arms: Patients undergoing noise cancellation during surgery
Procedure: Music is played but noise is not cancelled — In this group of patients, ambient noise cancelling was not applied and music, which has been proven to reduce anxiety in studies, was played during surgery.
  Arms: Patients who were played music during the operation

SUMMARY:
The aim of this clinical trial is to compare the effects of music and ambient noise cancellation during total knee arthroplasty and to analyse the effects on patients. The study will also collect information on patients' functional knee scores and anxiety levels. The main questions to be answered are the following:

Does the blocking of music or ambient noise, which is predicted to reduce anxiety, reduce people's anxiety levels? To what extent are participants affected by ambient noise? Does music or ambient noise blocking lead to an improvement in patients' functional scores?

The researchers will work with 3 groups of patients who will be exposed to ambient noise blocking, music playing and ambient noise during knee replacement surgery.

Participants will do the following:

Be asked questions about anxiety and knee function scores before and after surgery.

Attend clinical examinations at specified times for checks and tests. Outcomes will be assessed and recorded at appropriate times.

DETAILED DESCRIPTION:
Osteoarthritis is a degenerative and progressive knee disease that causes progressive loss of articular cartilage. According to the study by Harvey et al., osteoarthritis, the most common form of arthritis, is the most common cause of joint function limitation among the elderly. Osteoarthritis is common in load-bearing joints and one of these joints is the knee joint. According to a study by Dawson et al, the rate of symptomatic knee and hip osteoarthritis in individuals over 65 years of age was reported to be 40%. In patients with gonarthrosis (knee osteoarthritis), lifestyle changes, drug therapy and rehabilitation are recommended in the early stages (Stages 1-2), while total knee arthroplasty comes to the fore in the later stages (Stages 3-4).

Orthopaedic surgery operating rooms are generally known as noisy working environments. Especially joint surgeries such as total knee arthroplasty and total hip arthroplasty have a close relationship with noise due to the cutting motors, hammers and osteophyte excision procedures used during surgery. This noise during surgery may be associated with anxiety and delayed onset of movement in the postoperative period.

It is thought that the sympathetic nervous system, which is activated as a result of anxiety, may cause delayed wound healing and delay in the return of functional activity with the release of stress hormones. The use of music as a medical treatment has gained importance in recent years. According to the study of Wu et al. it was observed that music in the environment during awake craniotomy decreased anxiety, pulse rate and blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with stage 3-4 gonarthrosis
* Patients under spinal anaesthesia
* Patients undergoing unilateral knee replacement

Exclusion Criteria:

* Male patients
* Patients under 55 years of age
* Patients with a history of previous knee joint surgery
* Patients with a known history of rheumatological disease and inflammatory arthropathy
* Patients with dementia
* Patients with psychiatric illness
* Patients taking anxiolytic and antidepressant drugs without any history of psychiatric illness
* Patients with a history of active smoking
* Patients with hearing problems
* Illiterate patients
* Patients under general anaesthesia
* Patients with bilateral prosthesis

Min Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Knee Society Score Pre and Post-Operative | Pre-operative, Post-operative 3rd and 6th months
  Patients will be scored preoperatively and postoperatively by measuring the Knee Society Score. Maximum 100 points, the higher the score, the better the results.

SECONDARY OUTCOMES:
The Oxford Knee Score | Pre-operative, Post-operative 3rd and 6th months
  Patients will be scored preoperatively and postoperatively by measuring the The Oxford Knee Score. The Oxford Knee Score is frequently used to assess pain and functional limitations after knee arthroplasty, on a scale ranging from 0 to 48 (worst to best)
The Visual Analogue Scale | Postoperative 0-1-6-24-48-72 hours, 3rd week, 6th week, 3rd month, 6th month
  The pain Visual Analogue Scale is a unidimensional measure of pain intensity, used to record patients' pain progression, or compare pain severity between patients with similar conditions, on a scale ranging from 0 to 10. A score of 0 indicates no pain, a score of 10 indicates the worst pain
Short Form 36 | Preoperative, postoperative 6th month
  The Short Form 36 is a multipurpose, short-form health survey including 36 questions particularly useful for comparing general and specific populations rather than individuals, score ranging from 0 to 100. Higher scores indicate better health status.
State-trait anxiety inventory STAI FORM TX-1 | Pre-operative, Post-operative 1st day
  The State-Trait Anxiety Inventory (STAI) is a widely used measure of trait and state anxiety. It can be used in clinical settings to diagnose anxiety and differentiate it from depressive syndromes. We used the STAI-TX1 State-Trait scale in our study. Scores range from 20 to 80, with higher scores correlating with greater anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Güzelali Özdemir, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara City Hospital Bilkent, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tran BW, Nowrouz MY, Dhillon SK, Xie KK, Breslin KM, Golladay GJ. The Impact of Music and Noise-Cancellation on Sedation Requirements During Total Knee Replacement: A Randomized Controlled Trial. Geriatr Orthop Surg Rehabil. 2020 Mar 4;11:2151459320910844. doi: 10.1177/2151459320910844. eCollection 2020. PMID 32181048
- [Background] Skaugen P. Bacillus Calmette-Guerin therapy for bladder carcinoma in situ: use in a clinical setting. Urol Nurs. 1997 Jun;17(2):69-71. No abstract available. PMID 9239141
- [Background] Laine C, Markson LE, Fanning TR, Turner BJ. Relationship between ambulatory care accessibility and hospitalization for persons with advanced HIV disease. J Health Care Poor Underserved. 1999 Aug;10(3):313-27. doi: 10.1353/hpu.2010.0633. PMID 10436730
- [Background] Harvey WF, Hunter DJ. The role of analgesics and intra-articular injections in disease management. Rheum Dis Clin North Am. 2008 Aug;34(3):777-88. doi: 10.1016/j.rdc.2008.05.006. PMID 18687282
- [Background] Dawson J, Linsell L, Zondervan K, Rose P, Randall T, Carr A, Fitzpatrick R. Epidemiology of hip and knee pain and its impact on overall health status in older adults. Rheumatology (Oxford). 2004 Apr;43(4):497-504. doi: 10.1093/rheumatology/keh086. Epub 2004 Feb 3. PMID 14762225
- [Background] Wu PY, Huang ML, Lee WP, Wang C, Shih WM. Effects of music listening on anxiety and physiological responses in patients undergoing awake craniotomy. Complement Ther Med. 2017 Jun;32:56-60. doi: 10.1016/j.ctim.2017.03.007. Epub 2017 Mar 31. PMID 28619305